CLINICAL TRIAL: NCT02174965
Title: RSA-measured in Vivo Wear, Migration and Micromotion in the Corin Mini-Hip/Metafix and ECIMA Polyethylene.
Brief Title: Wear and Migration in the Corin Mini-Hip/Metafix and ECIMA Polyethylene
Acronym: MiniHip
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Oxford (Other)
Collaborators: Corin (Industry); Oxford University Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MiniHip
Record Dates: First submitted 2013-08-01; First posted 2014-06-26 (Estimated); Last update posted 2014-06-26 (Estimated); Status verified 2014-06

CONDITIONS: Hip Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Hip

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MiniHip (Corin U.K.) (Experimental): MiniHip (Corin U.K.) femoral component
  Interventions: Device: MiniHip (Corin U.K.)
- Metafix (Corin, U.K) (Active Comparator): Metafix (Corin, U.K) conventional cementless stem
  Interventions: Device: Metafix (Corin, U.K)

INTERVENTIONS:
Device: MiniHip (Corin U.K.) — MiniHip (Corin U.K.) femoral component
  Arms: MiniHip (Corin U.K.)
Device: Metafix (Corin, U.K) — Metafix (Corin, U.K) conventional cementless stem
  Arms: Metafix (Corin, U.K)

SUMMARY:
The primary objective of this study is to determine whether the Mini Hip (Corin, U.K.) femoral component has a predictable and stable migration pattern (mean migration of the femoral component in three-dimensions,in mm) over a three year period, compared to a conventional cementless stem (Metafix, Corin, U.K.). The secondary objectives of this study are to determine whether the Trinity (Corin, U.K.) acetabular component has a predictable and stable migration pattern over a three year period and to measure the linear wear of femoral head into the ECIMA Highly Cross-linked polyethylene.

ELIGIBILITY:
Inclusion Criteria:

* Women and men between the ages of 18 and 65 years old.
* Scheduled to receive a hip replacement
* Willing and able to give informed consent for participation in the study.
* Diagnosed with hip osteoarthritis
* Able (in the investigators opinion) and willing to comply with all study requirements.
* Willing to allow his/her General Practitioner and consultant, if appropriate, to be notified of participation in the study

Exclusion Criteria:

The participants may not enter the study if ANY of the following apply:

* Inflammatory arthropathy, osteoporosis or deformities of the proximal femur.
* Significant comorbidities that would make follow up difficult or uncomfortable
* Any other significant disease or disorder which, in the opinion of the investigator, may either put the participant at risk due to participation in the study, may influence the result of the study, or the participants ability to participate in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2012-09; Primary Completion 2022-09 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Radiostereometric Analysis (RSA) measured migration (mm) | Measured pre-operatively (baseline) and at 3, 6, 12, 18, 24 and 36 months post-operatively
  The images taken at each time point will be compared with the baseline to assess implant migration. Therefore the outcome is change in implant position measured using RSA.

SECONDARY OUTCOMES:
Dynamically Inducible Micromotion DIMM (mm) | Measured at 6, 12, 24 and 36 months post-operatively
  Using RSA this compares standard images with images taken in a single leg stance.
Implant failure for femoral and acetabular components | Observed at 3, 6, 12, 18, 24 and 36 months post-operatively
  Follow up assessment will monitor for signs of implant failure.
Change in Oxford Hip Score | Measured pre-operatively (baseline) and at 3, 6, 12, 18, 24 and 36 months post-operatively
  A PROM to assess patient benefit.
Change in Harris Hip Score | Measured pre-operatively (baseline) and at 3, 6, 12, 18, 24 and 36 months post-operatively
  A clinician recorded outcome score to assess functional improvement.

OTHER OUTCOMES:
DEXA Scan | Pre-operatively (baseline) and at 12 months post-operatively
  To monitor for peri-prosthetic changes in bone density following surgery

CONTACTS AND LOCATIONS:
Overall Officials: Sion Glyn-Jones, MA MBBS MRCS FRCS, Principal Investigator — University of Oxford
Locations (1):
- Nuffield Orthopaedic Centre, Oxford, United Kingdom